CLINICAL TRIAL: NCT02703753
Title: TOwards Prepared Mums (TOP-mums), for a Healthy Start: A Lifestyle Intervention to Reduce Overweight and Smoking in Women With a Pregnancy Wish to Prevent Perinatal Morbidity
Brief Title: TOP-mums, for a Healthy Start
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion was too slow, a lot of data loss during COVID pandemic
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: METC152026
Record Dates: First submitted 2016-02-25; First posted 2016-03-09 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Overweight; Obesity; Pregnancy Complications
MeSH Terms: conditions — Overweight; Obesity; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention is an integral and multidisciplinary lifestyle intervention consisting of a healthy diet, appropriate physical activity and, if applicable, smoking cessation, customised to the needs of the women.
  Interventions: Behavioral: Lifestyle intervention
- Control group (No Intervention): The control group will receive usual care, including standard lifestyle advices during consultation with the GP, midwife, obstetrician or at the child well being centre. Furthermore, the control group will receive 1 recipe for a healthy meal per week.

INTERVENTIONS:
Behavioral: Lifestyle intervention — The investigational treatment consists of a lifestyle intervention targeting on a healthy diet, physical activity and, if applicable, smoking cessation.
  Arms: Intervention group

SUMMARY:
This study evaluates the effect of a lifestyle intervention for women with a pregnancy wish who have a high risk on perinatal morbidity because of overweight or obesity. Half of the patients will receive the lifestyle intervention while the other half will receive usual care. It is hypothesized that an effective lifestyle intervention directed towards healthy living, including reduction of overweight or obesity and, if applicable, smoking reduction, health problems in mothers and their offspring can be prevented.

ELIGIBILITY:
Inclusion Criteria:

* Women with a pregnancy wish within 1 year;
* Aged 18-40 years;
* Overweight/obesity (BMI ≥ 25 kg/m2).

Exclusion Criteria:

* Haemodynamically significant heart disease;
* Restrictive lung disease;
* Congenital metabolic disease;
* Mentally retarded;
* Bariatric surgery;
* Diabetes type II, dependent on medicine.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Reduction in body weight | From baseline to 6 weeks postpartum

SECONDARY OUTCOMES:
Gestational weight gain | 6 weeks of gestational age to 36 weeks of gestational age
Postpartum weight retention | 6 weeks of gestational age to 6 months postpartum
Smoking cessation | Baseline. Prepregnancy: after 1, 2, 3, 6, 9 and 12 months. During pregnancy: at 6,12,20,32,36 and 40 weeks of gestational age. Postpartum: at 6 weeks and at 3, 6, 9 and 12 months.
Biochemical verification of tobacco use | Baseline. Prepregnancy: after 1, 2, 3, 6, 9 and 12 months. During pregnancy: at 6,12,20,32,36 and 40 weeks of gestational age. Postpartum: at 6 weeks and at 3, 6, 9 and 12 months.
  The amount of carbon monoxice (CO) in exhaled breath will be measured using a CO monitor (piCO Baby Smokerlyzer®, Bedfont, Kent, United Kingdom). Biochemical verification will also be done by measurement of urine cotinine.
Dietary habits | Baseline. Prepregnancy: after 3 and 12 months. During pregnancy: at 6 and 32 weeks of gestational age. Postpartum: 3 and 12 months.
  By a food diary and the three factor eating questionnaire.
Physical activity habits | Baseline. Prepregnancy: after 3 and 12 months. During pregnancy: at 6 and 32 weeks of gestational age. Postpartum: 3 and 12 months.
  By an accelerometer and the Baecke questionnaire.
Miscarriage | During pregnancy: at 6, 12 and 20 weeks of gestational age.
Time to pregnancy | From pregnancy wish to first day of last menstruation
Pregnancy complications | At birth
  Gestational diabetes mellitus, pregnancy-induced hypertension, preeclampsia.
Delivery complications | At birth
  Caesarean section, induction of labour, vacuum extraction, postpartum haemorrhage, maternal hospital stay, shoulder dystocia.
Vitamin D status | Will be measured at baseline and at 32 weeks of gestational age.
Dysmaturity and macrosomia | At birth
Prematurity | At birth
  Birth before 37 weeks of gestational age
Fasting glucose level | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
Fasting insulin level | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
Insuline resistance (HOMA-IR) | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
Total cholesterol | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
LDL cholesterol | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
HDL cholesterol | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
Triglycerides | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
Free fatty acids | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
Alkaline phosphatase | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
Gamma-GT | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
ASAT | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
ALAT | Will be measured at baseline; Prepregnancy: after 3 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: 3, 6 and 12 months.
Blood pressure | Will be measured at baseline; Prepregnancy: after 1, 2, 3, 6, 9 and 12 months; During pregnancy: at 6, 12, 20, 32, 36 and 40 weeks of gestational age; Postpartum: at 6 weeks and at 3, 6, 9 and 12 months.
Pulse wave velocity | Will be measured at baseline; Prepregnancy: after 3, 6 and 12 months; During pregnancy: at 6, 20 and 32 weeks of gestational age; Postpartum: at 6 and 12 months.
Fat mass and fatt free mass | Will be measured at baseline, at 32 weeks of gestational age during pregnancy and 6 months postpartum
  Body composition will be measured using the deuterium dilution method
Fasting glucose level of the child | At birth and 12 months postpartum
Fasting insulin level of the child | At birth and 12 months postpartum
Insulin resistance (HOMA-IR) of the child | At birth and 12 months postpartum
Total cholesterol of the child | At birth and 12 months postpartum
LDL cholesterol of the child | At birth and 12 months postpartum
HDL cholesterol of the child | At birth and 12 months postpartum
Triglycerides of the child | At birth and 12 months postpartum
Free fatty acids of the child | At birth and 12 months postpartum
Tidal volume of the child | Will be measured at 6 weeks and 12 months postpartum
Respiratory rate of the child | Will be measured at 6 weeks and 12 months postpartum
Respiratory system resistance of the child | Will be measured at 6 weeks and 12 months postpartum
Respiratory system reactance of the child | Will be measured at 6 weeks and 12 months postpartum
Endothelial vasodilatation of the child: Percentage change between baseline and maximum perfusion acetylcholine | Will be measured at 6 weeks and 3 and 12 months postpartum
Endothelial vasodilatation of the child: Percentage change between baseline and maximum perfusion nitroprusside | Will be measured at 6 weeks and 3 and 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Anita Vreugdenhil, MD, PhD, Principal Investigator — Maastricht UMC; Luc Zimmermann, Prof, MD, Study Chair — Maastricht UMC
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Timmermans YEG, van de Kant KDG, Reijnders D, Kleijkers LMP, Dompeling E, Kramer BW, Zimmermann LJI, Steegers-Theunissen RPM, Spaanderman MEA, Vreugdenhil ACE. Towards Prepared mums (TOP-mums) for a healthy start, a lifestyle intervention for women with overweight and a child wish: study protocol for a randomised controlled trial in the Netherlands. BMJ Open. 2019 Nov 19;9(11):e030236. doi: 10.1136/bmjopen-2019-030236. PMID 31748290